CLINICAL TRIAL: NCT04173429
Title: Efficacy and Safety of Nadroparin Calcium-Warfarin Sequential Anticoagulation in Portal Vein Thrombosis in Cirrhotic Patients：A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Anticoagulant Therapy in Portal Vein Thrombosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019126-QILU
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2017-01

CONDITIONS: Liver Cirrhosis; Portal Vein Thrombosis
Keywords: Portal vein thrombosis; Nadroparin calcium; Warfarin; Anticoagulation
MeSH Terms: conditions — Liver Cirrhosis | interventions — Nadroparin; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nadroparin calcium-warfarin sequential therapy group (Experimental): nadroparin calcium every 12 hours for 1 month followed by an oral administration of warfarin for 5 months
  Interventions: Drug: Nadroparin calcium, warfarin
- Control group (No Intervention): No anticoagulation therapy.

INTERVENTIONS:
Drug: Nadroparin calcium, warfarin — Nadroparin calcium subcutaneously every 12hs for 1 months followed by warfarin orally for 5 months. INR(international normalized ratio ) was detected every 3-4 days and adjusted carefully by 0.75mg dosage until achieve the target level of 2-3.
  Other Names: Experimental group
  Arms: nadroparin calcium-warfarin sequential therapy group

SUMMARY:
The study is aimed at evaluating the efficacy and safety of anticoagulant therapy with nadroparin calcium and warfarin in patients with portal vein thrombosis (PVT).

DETAILED DESCRIPTION:
Portal vein thrombosis (PVT) is a frequent complication of liver cirrhosis, referred to partial or complete thrombosis formed in the lumen of portal vein or/and branches of it. Currently, clinical guidelines of PVT in cirrhotic patients has not been addressed, and anticoagulant therapy of PVT patients with cirrhosis remains controversial. Although numerable studies have reported that anticoagulation therapy is effective, while a majority of them were respective and a few took control into consideration. In addition, no agreement has reached about the safety of anticoagulation. So, the efficacy and safety of anticoagulant therapy needs more prospective randomized controlled trial to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Liver cirrhosis diagnosis based on clinical, laboratory, and imaging studies, and PVT diagnosed by abdominal contrast-enhanced computed tomography, contrast-enhanced MRI, or portal angiography

Exclusion Criteria:

* Cavernous transformation of the portal vein
* Uncontrolled active bleeding
* Platelet count lower than 10*10^9/L
* Creatinine more than 170 mmol/L
* Ongoing or received antithrombotic/thrombolytic treatment
* Primary thrombophilia
* Budd-Chiari syndrome
* Pregnancy or breast-feeding period
* Severe cardiopulmonary diseases
* Severe systemic infection or sepsis
* Inability to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao, PhD.MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nadroparin Calcium-warfarin Sequential (NWS) Therapy Group: Nadroparin calcium every 12 hours for 1 month followed by an oral administration of warfarin for 5 months Nadroparin calcium, warfarin: Nadroparin calcium subcutaneously every 12hs for 1 months followed by warfarin orally for 5 months. INR(international normalized ratio ) was detected every 3-4 days and adjusted carefully by 0.75mg dosage until achieve the target level of 2-3.
Period: Overall Study
Arm/Group | Nadroparin Calcium-warfarin Sequential (NWS) Therapy Group | Control Group
Started | 32 | 32
Completed the Nadroparin Calcium Therapy and Received Warfarin | 32 | 0
Completed | 30 | 30
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Nadroparin Calcium-warfarin Sequential (NWS) Therapy Group: Nadroparin calcium every 12 hours for 1 month followed by an oral administration of warfarin for 5 months.
  Nadroparin calciumsubcutaneously every 12hs for 1 months followed by warfarin orally for 5 months. INR(international normalized ratio ) was detected every 3-4 days and adjusted carefully by 0.75mg dosage until achieve the target level of 2-3.
- Total: Total of all reporting groups
Arm/Group | Nadroparin Calcium-warfarin Sequential (NWS) Therapy Group | Control Group | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: year] — The minimum and maximum age of the participants was 18 and 75, respectively.
  year | 55 (9) | 53 (10) | 54 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 21 | 21 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Etiology [Count of Participants; unit: Participants]
  Hepatitis B virus (HBV) | 23 | 23 | 46
  Hepatitis C virus (HCV) | 0 | 1 | 1
  Alcoholic | 5 | 3 | 8
  Cryptogenic | 4 | 5 | 9
Child-Pugh score [Mean (Standard Deviation); unit: units on a scale] — The Child-Pugh score was an quantitative assessment of the liver function reserves. The five indexes including general situation, ascites, the concentration of serum bilirubin, serum albumin and prothrombin time were evaluated to calculate a score. The minimum and maximum Child-Pugh score was 5 and 15, respectively. The lower score indicated a better outcome.
  units on a scale | 6.51 (1.27) | 6.81 (1.44) | 6.59 (1.35)
Model for end-stage liver disease (MELD) score [Mean (Standard Deviation); unit: units on a scale] — The minimum and maximum MELD score was 0 and 18, respectively. A lower value was considered to be a better outcome.
  units on a scale | 9.13 (3.39) | 10.00 (3.65) | 9.51 (3.50)
Total bilirubin (μmol/L) [Mean (Standard Deviation); unit: μmol/L] — The Total bilirubin referred to the total bilirubine, including direct bilirubine and indirect bilirubine. The minimum and maximum value of Total bilirubin was 5 and 21umol/L, respectively.
  μmol/L | 18.64 (9.76) | 22.31 (17.00) | 20.3 (13.6)
Creatinine (μmol/L) [Mean (Standard Deviation); unit: μmol/L] — The minimum and maximum value of Creatinine was 62 and 115μmol/L, respectively.
  μmol/L | 60.90 (16.00) | 65.78 (16.07) | 63.2 (16.1)
International normalized ratio (INR) [Mean (Standard Deviation); unit: ratio] — The minimum and maximum value of INR was 0.8 and 1.2, respectively.
  ratio | 1.34 (0.23) | 1.36 (0.20) | 1.35 (0.21)
Platelet (*10^9 cells/L) [Mean (Standard Deviation); unit: *10^9 cells/L] — The minimum and maximum value of Platelet was 125 and 350*10^9 cells/L, respectively.
  *10^9 cells/L | 126.22 (170.86) | 134.63 (137.48) | 130 (150)
D-dimer(μg/mL) [Mean (Standard Deviation); unit: μg/mL] — The maximum value of D-dimer was 0.5μg/mL.
  μg/mL | 1.14 (1.05) | 1.50 (1.32) | 1.31 (1.19)
Albumin (g/L) [Mean (Standard Deviation); unit: g/L] — The minimum and maximum value of Albumin was 40 and 55g/L, respectively.
  g/L | 36.14 (5.25) | 35.03 (4.45) | 35.64 (4.89)
Low-density lipoprotein cholesterol(LDL-C,mmol/L) [Mean (Standard Deviation); unit: mmol/L] — The minimum and maximum value of Low-density lipoprotein cholesterol was 1.00 and 3.37mmol/L, respectively.
  mmol/L | 1.91 (0.69) | 1.77 (0.68) | 1.85 (0.68)
Triglyceride (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — The minimum and maximum value of Triglyceride was 0.3 and 1.7mmol/L, respectively.
  mmol/L | 0.95 (0.51) | 0.83 (0.36) | 0.89 (0.44)
Cholesterol (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — The minimum and maximum value of Cholesterol was 2.8 and 6.0mmol/L, respectively.
  mmol/L | 3.47 (1.02) | 3.50 (1.10) | 3.48 (1.05)
Esophageal varices [Count of Participants; unit: Participants]
  Yes | 26 | 27 | 53
  No | 6 | 5 | 11
Ascites [Count of Participants; unit: Participants]
  Yes | 17 | 20 | 37
  No | 15 | 12 | 27
Endoscopic treatment [Count of Participants; unit: Participants]
  Yes | 13 | 9 | 22
  No | 19 | 23 | 42
Splenectomy/Partial splenic embolization(PSE) [Count of Participants; unit: Participants]
  Yes | 9 | 13 | 22
  No | 23 | 19 | 42
Extent of portal vein thrombosis(PVT) [Count of Participants; unit: Participants]
  Main portal vein(MPV) only | 12 | 14 | 26
  Superior mesenteric vein(SMV) only | 2 | 3 | 5
  Splenic vein(SV) only | 0 | 2 | 2
  MPV + SMV | 17 | 9 | 26
  MPV + SV | 0 | 2 | 2
  MPV + SMV + SV | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Recanalization Rate
Description: For each venous segment, the vein and residual patent lumen were outlined at the level of the maximum thrombosis. Total lumen area and patent lumen area were calculated with commercially available software. The degree of thrombus occlusion was estimated as a percentage by thrombosis area/total lumen area×100%. The primary outcome was the overall recanalization rate, both complete and partial. Complete recanalization was referred to the complete disappearance of the thrombus in the portal vein trunk, at least one of the two intrahepatic portal vein branches, SMV and SV. Partial recanalization was defined as a more than 50% reduction of the thrombus, with the thrombus not extending to other veins.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Nadroparin Calcium-warfarin Sequential Therapy Group: nadroparin calcium every 12 hours for 1 month followed by an oral administration of warfarin for 5 months
  Low molecular weight heparin (LMWH), warfarin: Low molecular weight heparin subcutaneously every 12hs for 1 months followed by warfarin orally for 5 months(LMWH-warfarin group). INR(international normalized ratio ) was detected every 3-4 days and adjusted carefully by 0.75mg dosage until achieve the target level of 2-3.
Arm/Group | Nadroparin Calcium-warfarin Sequential Therapy Group | Control Group
Number analyzed (Participants) | 32 | 32
Participants | 20 | 11

2. Secondary Outcome: Rate of Bleeding
Description: Risk of bleeding episodes
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nadroparin Calcium-warfarin Sequential (NWS) Therapy Group | Control Group
Number analyzed (Participants) | 32 | 32
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Nadroparin Calcium-warfarin Sequential (NWS) Therapy Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 1/32 | 0/32
OTHER ADVERSE EVENTS (reported when occurring in more than 3.12% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nadroparin Calcium-warfarin Sequential (NWS) Therapy Group (N=32) | Control Group (N=32)
Bleeding events (Gastrointestinal disorders) | 1 | 0 — Bleeding events consisted of hematemesis, melena, epistaxis, injection-site hemorrhage, and other bleeding events. One patient in the NWS therapy group experienced hematemesis during warfarin administration and discontinued the therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04173429/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04173429/SAP_001.pdf